CLINICAL TRIAL: NCT01198535
Title: Phase I Study of Cetuximab With RO4929097 in Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02905; NCI-2012-02905 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICC GI 09106 (Other: Vanderbilt University/Ingram Cancer Center); 8511 (Other: CTEP); N01CM00100 (NIH); P30CA068485 (NIH); NCT01207882 (obsolete NCT alias)
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2012-12

CONDITIONS: Colon Mucinous Adenocarcinoma; Colon Signet Ring Cell Adenocarcinoma; Rectal Mucinous Adenocarcinoma; Rectal Signet Ring Cell Adenocarcinoma; Recurrent Colon Carcinoma; Recurrent Rectal Carcinoma; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide

ARMS (2):
- Arm A (RO4929097, cetuximab) (Experimental): Patients in Arm A will receive cetuximab at the standard dose: 400 mg/m2 IV loading dose on Day 1 followed by cetuximab 250 mg/m2 IV weekly. The RO4929097 will be dose escalated starting at 20 mg given daily 3 days on, 4 days off, weekly. The dose levels of RO4929097 to be explored will be 20 mg, 30 mg, 45 mg, 90 mg, 140 mg given days 1-3 weekly. No intrapatient dose escalation will be allowed.
  Interventions: Biological: Cetuximab; Drug: Gamma-Secretase Inhibitor RO4929097; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Arm B (RO4929097, cetuximab) (Experimental): Patients in Arm B will receive cetuximab 200 mg/m2 IV weekly without a loading dose. The RO4929097 will be dose escalated starting at 20 mg given daily 3 days on, 4 days off, weekly. The dose levels of RO4929097 to be explored will be 20 mg, 30 mg, 45 mg, 90 mg, 140 mg given days 1-3 weekly. No intrapatient dose escalation will be allowed.
  Interventions: Biological: Cetuximab; Drug: Gamma-Secretase Inhibitor RO4929097; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
Drug: Gamma-Secretase Inhibitor RO4929097 — Given PO
  Other Names: RO4929097
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
The purpose of this study is to determine if a new drug, RO4929097, can work with cetuximab, a drug already approved for colorectal cancer, to help fight the patient's cancer. Cancers arise as a result of abnormal control of gene expression. One of the pathways that gets abnormally regulated in some cancers is the Notch pathway. RO4929097 is an investigational drug that blocks the activation of the Notch pathway. It is hoped that by blocking this abnormal activation, this drug may be helpful in patients with cancer but the investigators do not yet know if that is true. Cetuximab is an antibody against epidermal growth factor receptor and is known to have activity in metastatic colorectal cancer. Recent studies have shown that people with colorectal cancers that contain a mutation in a gene called K-ras do not benefit from receiving cetuximab. It is unknown if adding RO4929097 to cetuximab would benefit patients who have tumors with this mutation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determination of the maximum tolerated dose (MTD) of the combination of cetuximab and RO4929097.

SECONDARY OBJECTIVES:

I. Safety and tolerability of the combination of cetuximab and RO4929097. II. Exploratory analyses of anti-tumor effect with the combination. III. Laboratory correlatives exploring response rate with notch receptors and ligand expression, correlation of response and toxicity profiles to expression of EGFR pathway components, and evaluation of serum and tissue markers of gamma-secretase inhibitor activity.

IV. Pharmacokinetic studies.

OUTLINE: This is a dose-escalation study of gamma-secretase/Notch signalling pathway inhibitor RO4929097.

Phase I dose escalation: In this part of the study, the investigators are trying to find out what is the highest tolerated dose of RO4929097 that can be safely combined with cetuximab. The investigators will be testing two different cetuximab doses. One is the standard dose (Arm A) and one is a little less than the standard dose (Arm B). Everyone will get treated with cetuximab and R04929097 in this part of the study.

Phase I dose expansion: In this part of the study, the investigators will take the highest tolerated dose found in the phase I part of the study and test a small number of people with colorectal cancer to see if there is any activity with the combination of drugs. Everyone will get treated with cetuximab and RO4929097 in this part of the study. This part of the study will be restricted to patients whose tumors do not have a mutation in the K-ras gene. RO4929097 is an investigational anti-cancer agent that has not yet been approved by the Food and Drug Administration (FDA) for use in colorectal cancer. Cetuximab is FDA approved for metastatic colorectal cancer.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic colorectal adenocarcinoma
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Patients must have received at least one prior therapy for metastatic disease; prior therapy with anti-EGFR antibody is allowed only as long as patient did not require dose reductions of the anti-EGFR antibody because of poor tolerability
* Life expectancy of greater than 3 months
* ECOG performance status =<2 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin within normal institutional limits if no liver metastases
* Total bilirubin < 1.5 X the institutional upper limit of normal if liver metastases are present
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal if no liver metastases
* AST(SGOT)/ALT(SGPT) < 5 X institutional upper limit of normal if liver metastases are present
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* For the phase I dose expansion, tumor must be KRAS wildtype
* There must be available a tumor block or 20 unstained slides for correlative studies
* The effects of RO4929097on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because Notch signal pathway inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of childbearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, for the duration of study participation, and for at least 12 months post-treatment; should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study and for 12 months after study participation, the patient should inform the treating physician immediately

  * Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 10-14 days and within 24 hours prior to the first dose of RO4929097 (serum or urine); a pregnancy test (serum or urine) will be administered every 4 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of RO4929097; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing RO4929097, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of RO4929097
  * Female patients of childbearing potential are defined as follows:

    * Patients with regular menses
    * Patients, after menarche with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
    * Women who have had tubal ligation
  * Female patients may be considered to NOT be of childbearing potential for the following reasons:

    * The patient has undergone total abdominal hysterectomy with bilateral salpingo-oophorectomy or bilateral oophorectomy
    * The patient is medically confirmed to be menopausal (no menstrual period) for 24 consecutive months
* Ability to understand and the willingness to sign a written informed consent document
* Ability to swallow pills

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered to a grade 1 or less from adverse events due to agents administered more than 4 weeks earlier with the exception of alopecia and neuropathy
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to RO4929097 or other agents (EGFR antibodies) used in the study
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®) are ineligible
* Preclinical studies indicate that RO4929097 is a substrate of CYP3A4 and inducer of CYP3A4 enzyme activity. Caution should be exercised when dosing RO4929097 concurrently with CYP3A4 substrates, inducers, and/or inhibitors; furthermore, patients who are taking concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4 should be switched to alternative medications to minimize any potential risk; if such patients cannot be switched to alternative medications, they will be ineligible to participate in this study
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption; patients must be able to swallow tablets
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, a history of torsades de pointes, significant cardiac arrhythmia other than chronic, stable atrial fibrillation, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because RO4929097 is a Notch pathway inhibiting agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with RO4929097, breastfeeding should be discontinued if the mother is treated with RO4929097; these potential risks may also apply to other agents used in this study
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with RO4929097; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy
* Cardiovascular: baseline QTcF > 450 msec (male) or QTcF > 470 msec (female)
* Patients whose tumor contains a mutation in KRAS are not eligible for the phase I dose expansion portion of the study
* Patients with prior exposure to γ-secretase inhibitors
* Patients with another active malignancy
* Patients on antiarrhythmics or other medications known to prolong QTc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
MTD of RO4929097 | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Emily Chan, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States